CLINICAL TRIAL: NCT03424369
Title: Correlation Analysis Between Eustachian Tube Function and Prognosis of Tympanoplasty
Brief Title: Correlation Analysis Between ETF and Prognosis of Tympanoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ETF and tympanoplasty
Record Dates: First submitted 2018-01-16; First posted 2018-02-07 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Eustachian Tube Dysfunction
MeSH Terms: interventions — Tympanoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eustachian tube unobstructed
  Interventions: Procedure: Tympanoplasty
- Eustachian tube dysfunction
  Interventions: Procedure: Tympanoplasty

INTERVENTIONS:
Procedure: Tympanoplasty — Tympanoplasty

SUMMARY:
The regular opening of the eustachian tube plays an important role in maintaining normal pressure in middle ear cavity, hearing function and preventing the occurrence of middle ear inflammation. The current evaluation of Eustachian tube function mainly depends on the patient's history of auricular distention, occlusion, physical examination (Valsalva), acoustic impedance test. However, these tests can not accurately assess the eustachian tube function, the lack of quantitative analysis of eustachian tube function. Currently, surgical treatment of patients with chronic otitis media is one of the most important treatment methods. However, the current results show that some patients can not reconstruct the gas-containing structure of the middle ear after operation, which brings about the treatment of diseases and the recovery of auditory function Difficulties. Although domestic and foreign scholars believe that eustachian tube function in tympanoplasty in the reconstruction of the middle ear with air cavity plays an important role, but due to the lack of a reliable quantitative evaluation of eustachian tube function, eustachian tube function in the occurrence of chronic otitis media , There is a lack of reliable evidence-based medicine in the assessment of the value of development and prognosis. In recent years, a new eustachian tube function evaluation method - Eustachian tube manometry technique, began a quantitative objective assessment of Eustachian tube function, combined with physical examination and subjective symptom scales to conduct a comprehensive assessment of eustachian tube function . This study wants to evaluate the eustachian tube function preoperatively and postoperatively in patients with chronic otitis media who underwent surgery. Regular postoperative follow-ups were used to understand the importance of eustachian tube function in the prognosis of chronic otitis media surgery , In order to further improve the eustachian tube function and improve the surgical curative effect of chronic otitis media.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years old, gender is not limited; 2.clear diagnosis of chronic otitis media, middle ear cholesteatoma need tympanoplasty patients; 3.Subjects or their legal representatives can understand the purpose of the study, show sufficient compliance with the research protocol, and sign the informed consent form.

Exclusion Criteria:

1. secondary chronic otitis media (after head and neck cancer radiotherapy);
2. ipsilateral ear recurrence after surgical treatment, requiring secondary surgery;
3. two tympanoplasty surgery;
4. typical allergic rhinitis, nasal endoscopy or imaging studies suggest chronic rhinosinusitis, nasal polyps and other short-term eustachian tube function of a greater impact on the disease;
5. poor general health, with severe liver and kidney dysfunction, coagulation disorders, cardiovascular disease, neurological diseases can not tolerate surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the results of Eustachian tube manometry, the patients were divided into two groups: Eustachian tube function state and Eustachian tube dysfunction group. The prognosis of tympanoplasty was compared, and the eustachian tube function state was defined in tympanic cavity of chronic otitis media The value of postoperative recovery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Eustachian tube function status were evaluated using TUBOMANOMETRY (TMM) | before the surgery, and 6months after the surgery
  Eustachian tube functional status in patients with chronic otitis media before/after tympanoplasty were evaluated using TUBOMANOMETRY (TMM)

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No